CLINICAL TRIAL: NCT05683808
Title: Venous Thromboembolism Prevention in Outpatients With Glioma
Acronym: VTE-POG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); MaineHealth (Other)
Responsible Party: Principal Investigator, Alissa Thomas, Associate Professor of Neurological Sciences, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NNECOS004
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma; Astrocytoma; Venous Thromboembolism
Keywords: High grade glioma; Glioblastoma; Astrocytoma; Venous thromboembolism; Apixaban
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Venous Thromboembolism; Glioma | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Open label study of apixaban for VTE prevention in patients with newly diagnosed grade 4 glioma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm study (Experimental)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Open label

SUMMARY:
This is an open label study of apixaban for venous thromboembolism prevention in patients with newly diagnosed grade 4 glioma.

DETAILED DESCRIPTION:
Patients with primary brain tumors, including glioblastoma and astrocytoma, are at high risk of developing venous thromboemboli (VTE) as a comorbid condition. Prior studies have demonstrated safety and efficacy of primary pharmacological prevention of VTE using blood thinning medications, including apixaban. These studies have included a small cohort of patients with grade 4 glioma. The purpose of this study is to gather additional safety data regarding the use of apixaban for primary prevention of VTE in patients with newly diagnosed grade 4 glioma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of malignant glioma, World Health Organization (WHO) grade 4, including glioblastoma and astrocytoma, based on recent biopsy or resection.
* Age 18 and old
* Karnofsky performance status (KPS) 60-100
* Acceptable labs, including platelets of greater than or equal to 100,000, glomerular filtration rate (GFR) greater than or equal to 25.
* Ability to provide informed consent.
* Planning for treatment with radiation and chemotherapy.

Exclusion Criteria:

* Evidence of deep venous thrombosis (DVT), pulmonary embolism (PE), or cerebral vein thrombosis (CVT) within 6 months prior to enrollment on the study.
* Pregnancy.
* Significant bleeding risk including: history of symptomatic intracranial hemorrhage, active bleeding at time of study registration, clinically significant bleeding within 14 days of study registration, intracranial trauma in the past 6 months, including stroke or traumatic brain injury, major surgery or major procedure within 48 hours.
* Allergy to apixaban or contraindication to prophylactic anticoagulation. Contraindications include patients who are currently on unfractionated heparin, low molecular weight heparin, heparin derivatives (examples: fondaparinux), or other direct oral anticoagulants (examples: dabigatran, edoxaban, rivaroxaban), who are either unable or unable to discontinue these agents in favor of the investigational drug. Apixaban is also contraindicated in patients who are on strong CYP3A4 inhibitor and P-glycoprotein inhibitors.
* Indication for full anticoagulation (i.e. atrial fibrillation, mechanical valve, etc.).
* Estimated life expectancy of <3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of apixaban as determined by bleeding risk | 6 months
  CTCAE 5 reporting of grade 2 non-Central Nervous System (CNS) hemorrhage or grade 2 new CNS hemorrhage.

SECONDARY OUTCOMES:
Efficacy in prevention of venous thromboembolism | 6 months
  Incidence of VTE

CONTACTS AND LOCATIONS:
Overall Officials: Alissa A Thomas, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States